CLINICAL TRIAL: NCT05940142
Title: Prediction of Propofol Effect Compartment Concentrations
Acronym: Propo2022
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Karl Landsteiner University of Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: SF44
Record Dates: First submitted 2023-05-14; First posted 2023-07-11 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-05

CONDITIONS: Analysis of Anaesthesia Depth

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn about the prediction of the effect of Propofol by means of EEGs. The main questions it aims to answer are:

* Develop models that can reliably predict the effect of Propofol
* Select the most well suited model for clinical practice
* Compare this model to already existing models (e.g. Schnider-model)

Participants will asked to allow us to collect and use the EEG data recorded during the operations.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 or older at the time of the signature of the informed consent
* Signed informed consents
* Planned TIVA with Propofol

Exclusion Criteria:

* Use of extracorporal circulation (e.g., HLM, ECMO)
* Admission to an ICU/IMCU before the operation or planned admission to an ICU/IMCU after the operation
* Administration of Propofol seven days prior to the planned operation
* Missing informed consent
* All contraindications against TIVA (e.g., allergy against Propofol or soy)
* All operations where BIS monitoring cannot be used (e.g., skin lesions on the front)
* Patients for which the administration of Propofol could be potentially harmfull (e.g., severe heart failure with the risk of drop of blood pressure)
* Neurosurgical operations

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients meeting the inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Bilateral BIS values (derived from EEG) | During procedure (From the beginning of general anaesthesia (induction of anaesthesia) until the patient has woken up (end of anaesthesia)).
  Comparison of Predicted and Measured EEG values (recorded every five seconds)
Propofol cumulative dose | During procedure (From the beginning of general anaesthesia (induction of anaesthesia) until the patient has woken up (end of anaesthesia)).
  Cumulative dose of Propofol (recorded every second)

CONTACTS AND LOCATIONS:
Locations (1):
- Klinische Abteilung für Anästhesie und Intensivmedizin, Krems, Lower Austria, Austria